CLINICAL TRIAL: NCT03732443
Title: Translation and Validation of the Family Confusion Assessment Method (FAM-CAM) Into German for the Detection of Delirium in Critically Ill Patients
Brief Title: FAM-CAM Translation and Validation Into German
Acronym: TRAVAGE-FAM
Status: Withdrawn | Type: Observational
Why Stopped: Errors in study conception, e.g. sample size calculation.
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: TRAVAGE-FAM
Record Dates: First submitted 2018-10-29; First posted 2018-11-06 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Delirium; Critical Illness; Family Members
Keywords: Delirium; Family Members; Critical Illness; ABCDEF; Validation; Translation; FAMCAM; CAM-ICU
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical Ill Patients: Critically ill patients with a RASS ≥ 3. FAM-CAM and CAM-ICU will be administered.
  Interventions: Diagnostic Test: FAM-CAM

INTERVENTIONS:
Diagnostic Test: FAM-CAM — Family Confusion Assessment Method

SUMMARY:
Validation and Translation of the Family Confusion Assessment Method (FAM-CAM) into German according to Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes of the International Society for Pharmaoeconomics and Outcome Research and comparison to CAM-ICU.

ELIGIBILITY:
Inclusion Criteria:

* Intensive Care Stay ≥ 48 hours
* Expected RASS ≥ 3
* Communication possible in German (minimum of C1 level of Common European Framework of Reference for Languages)

Exclusion Criteria:

* preexisting psychosis, dementia or depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients which are at risk for delirium and where assessing of delirium is not limited by language barriers.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Cohen's Kappa Coefficient | During a family visit which is not the first while treated in intensive care (an median of 10 days)
  Cohen's Kappa coefficient comparing the Family Confusion Assessment Method and the Confusion Assessment Method for Intensive Care Unit

SECONDARY OUTCOMES:
Specificity of FAM-CAM | During a family visit which is not the first while treated in intensive care (an median of 10 days)
  Specificity of the Family Confusion Assessment Method in critically ill patients to detect Delirium
Sensitivity of FAM-CAM | During a family visit which is not the first while treated in intensive care (an median of 10 days)
  Sensitivity of the Family Confusion Assessment Method in critically ill patients to detect Delirium
NPV of FAM-CAM | During a family visit which is not the first while treated in intensive care (an median of 10 days)
  Negative Predictive Value of the Family Confusion Assessment Method in critically ill patients to detect Delirium
PPV of FAM-CAM | During a family visit which is not the first while treated in intensive care (an median of 10 days)
  Positive Predictive Value of the Family Confusion Assessment Method in critically ill patients to detect Delirium

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Klinikum rechts der Isar der TUM
Locations (1):
- Klinikum rechts der Isar der TUM, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing can be requested for research collaboration purpose or meta-analysis. A data share agreement will have to be signed.

REFERENCES:
- [Background] Flanagan NM, Spencer G. Informal caregivers and detection of delirium in postacute care: a correlational study of the confusion assessment method (CAM), confusion assessment method-family assessment method (CAM-FAM) and DSM-IV criteria. Int J Older People Nurs. 2016 Sep;11(3):176-83. doi: 10.1111/opn.12106. Epub 2015 Dec 16. PMID 26669904
- [Background] Aya AGM, Pouchain PH, Thomas H, Ripart J, Cuvillon P. Incidence of postoperative delirium in elderly ambulatory patients: A prospective evaluation using the FAM-CAM instrument. J Clin Anesth. 2019 Mar;53:35-38. doi: 10.1016/j.jclinane.2018.09.034. Epub 2018 Oct 4. PMID 30292069
- [Background] Steis MR, Evans L, Hirschman KB, Hanlon A, Fick DM, Flanagan N, Inouye SK. Screening for delirium using family caregivers: convergent validity of the Family Confusion Assessment Method and interviewer-rated Confusion Assessment Method. J Am Geriatr Soc. 2012 Nov;60(11):2121-6. doi: 10.1111/j.1532-5415.2012.04200.x. Epub 2012 Oct 5. PMID 23039310